CLINICAL TRIAL: NCT03202004
Title: A Double-Blind Safety and Efficacy Study of GSK2894512 Cream Versus Vehicle in the Treatment of Adult Plaque Psoriasis
Brief Title: GSK2894512 Vehicle-Controlled Study for Adult Plaque Psoriasis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision not to progress the planned Phase 3 studies is a business decision based on the need to prioritise and focus resources within GSK.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry); ERT: Clinical Trial Technology Solutions (Other); Q2 Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200852
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Psoriasis
Keywords: PGA; efficacy; PASI; GSK2894512; NRS; Topical; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator, study center staff, subject, and sponsor will be blinded to randomized study treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK2894512 1% cream group (Experimental): Subjects will apply a thin layer of GSK2894512 1% (10 milligrams per gram [mg/g]) topical cream once daily to all psoriasis lesions for 12 weeks. The study staff will instruct subjects on proper topical application of cream.
  Interventions: Drug: GSK2894512 1% cream
- Vehicle cream group (Placebo Comparator): Subjects will apply a thin layer of vehicle cream once daily to all psoriasis lesions for 12 weeks. The study staff will instruct subjects on proper topical application of cream.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: GSK2894512 1% cream — 1 % (10 mg/g) GSK2894512 cream will be provided in tubes labeled in compliance with country requirements.
  Arms: GSK2894512 1% cream group
Drug: Vehicle cream — Vehicle cream will be provided in tubes labeled in compliance with country requirements.
  Arms: Vehicle cream group

SUMMARY:
This study will evaluate the efficacy and safety of GSK2894512 cream for the topical treatment of plaque psoriasis (psoriasis) with its vehicle cream. This is a randomized, double-blind, vehicle-controlled, parallel-group, multicenter study in adults with psoriasis. The aim of this study is to show superiority of GSK2894512 over vehicle by comparing their response rates. The study will consist of 3 periods: up to 4 weeks screening, 12 weeks blinded treatment, and 1 week post-treatment follow-up period. Subjects will apply randomized study treatment to all psoriasis lesions once daily for 12 weeks. Subjects will be stratified by Baseline physician global assessment (PGA) category (PGA score=2, PGA score >=3) at randomization. Approximately 120 subjects will be randomized into the study of which 80 will receive GSK2894512 1% cream and 40 will receive vehicle cream. Total duration of a subject's participation in the study will be approximately for 14 to 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years at the time of signing the informed consent.
* Clinical diagnosis of chronic stable plaque psoriasis. Diagnosis and chronicity to be confirmed and documented by an experienced dermatologist.
* Body surface area involvement >=2%.
* A PGA score of >=2.
* One target plaque located on the trunk or extremities that is at least 9 centimeter (cm)^2 in size with a target plaque severity score (TPSS) >=5 and an induration sub score >=2. Primary target plaque should not be located on the knees, elbows, feet, ankle, hands, intertriginous areas, face, or scalp.)
* Male or female. A female is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * Is a WOCBP who agrees to follow the specified contraceptive guidance throughout the study, including screening, during the treatment period, and for at least 1 week after the last exposure to study treatment.
* Capable of giving signed informed consent

Exclusion Criteria:

* Psoriasis other than plaque variant.
* Any sign of infection of any of the psoriatic lesions.
* Concurrent conditions and history of other diseases:

  * Immunocompromised (examples: lymphoma, acquired immunodeficiency syndrome) or have a history of malignant disease within 5 years before the Baseline visit.
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before the Baseline visit.
  * Active acute bacterial, fungal, or viral (examples: herpes simplex, herpes zoster, chicken pox) skin infection within 1 week before the Baseline visit
  * Significant dermatologic or inflammatory condition other than plaque psoriasis that, in the investigator's opinion, would make it difficult to interpret data or assessments during the study.
* A history or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* Known hypersensitivity to GSK2894512 or excipients of the study treatments, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation.
* Alanine transferase (ALT) >2 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Stable chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C, examples: presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody test result at screening or within 3 months prior to starting study treatment) is acceptable if the subject otherwise meets entry criteria.
* QT interval corrected for heart rate according to Fridericia's formula QTcF >450 milliseconds (msec) or QTcF >480 msec in subjects with bundle branch block.
* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation (examples: phototherapy, tanning beds/booths, or therapeutic sunbathing) within 4 weeks prior to the Baseline visit and/or intention to have such exposure during the study, which could potentially impact the subject's psoriasis (as determined by the investigator).
* Used any of the following treatments within the indicated period before the Baseline visit:

  * Minimum of 5 half-lives for biologic agents -12 months: rituximab or efalizumab; 8 months: ustekinumab; 5 months: secukinumab; 12 weeks: golimumab; 10 weeks: ixekizumab; 8 weeks: infliximab, adalimumab, or alefacept; 4 weeks: etanercept (list is not exclusive, contact medical monitor for questions).
  * 4 weeks -systemic treatments: cyclosporin, interferon, methotrexate, apremilast, tofacitinib, mycophenolate, thioguanine, hydroxyurea, sirolimus, azathioprine, other systemic immunosuppressive or immunomodulating agents, fumaric acid derivatives, vitamin D3 and analogs, retinoids (examples: acitretin, isotretinoin), psoralens, corticosteroids, or adrenocorticotropic hormone analogs.
  * 2 weeks -immunizations; drugs known to possibly worsen psoriasis, such as beta-blockers (example, propranolol), lithium, iodides, angiotensin-converting enzyme inhibitors, and indomethacin, unless on a stable dose for >12 weeks.
  * 2 weeks -topical treatments: corticosteroids, immunomodulators, anthralin (dithranol), Vitamin D derivatives (examples: calcipotriene, calcipotriol), retinoids (example, tazarotene), or coal tar (used on the body).
* Participated in a clinical study and received an investigational product within the following time period prior to the Baseline visit: 4 weeks, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participated in a previous study using GSK2894512 or WBI-1001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-22 (Estimated); Primary Completion 2018-09-28 (Estimated); Study Completion 2018-09-28 (Estimated)

PRIMARY OUTCOMES:
Proportion OF SUBJECTS WITH PGA SCORE OF CLEAR OR ALMOST CLEAR (0 OR 1) AND A MINIMUM 2-GRADE IMPROVEMENT IN PGA SCORE FROM BASELINE AND WEEK 12 | Baseline (Day 1) and Week 12
  PGA is a clinical tool (a 5 point scale) for assessing the current state/severity of a subject's psoriasis. It is a morphological assessment of overall disease severity, as determined by the investigator, using the clinical characteristics of erythema, scaling, and plaque thickness/elevation as guidelines. Subjects will be scored using the following categories: 0=Clear; 1=Almost clear; 2=Mild; 3=Moderate; and 4=Severe.

SECONDARY OUTCOMES:
Proportion of subjects with >=75% improvement in Psoriasis Area and Severity Index (PASI) from Baseline to Week 12 | Baseline (Day 1) and up to Week 12
  The PASI scoring system is a widely-used standard clinical tool for assessing the severity of psoriasis that takes into account the overall severity of erythema (redness), induration (plaque thickness), and scale, and the extent of percent body surface area (%BSA) affected with psoriasis. The 3 clinical signs are each graded on a 5-point scale (0=None; 4=Severe) and the % BSA affected is scored on a 7-point scale (0=0%; 6>=90%) for each of the 4 specified body regions (head, upper extremities, trunk, and lower extremities). The individual scores are multiplied by a weighted factor for each body region; the sum of these scores gives the overall PASI score. Higher scores indicate more severe disease.
Proportion OF SUBJECTS WITH>=3-POINT REDUCTION IN WEEKLY AVERAGE ITCH/PRURITUS NUMERIC RATING SCALE (NRS) FROM BASELINE TO WEEK 12 FOR SUBJECTS WITH A BASELINE SCORE >=4 | Baseline (Day 1) and up to Week 12
  The severity and bother of psoriasis-related itching, stinging, burning, pain, and scaling and impact items about the embarrassment, avoidance of activities with other people, and movement restrictions will be assessed using Psoriasis Symptom Diary. It is a 16-item electronic, daily (24-hour recall), validated assessment that measures self-reports of psoriasis symptoms and impact on functional health. Each item will be rated on a 0 to 10 NRS, with unlabeled numbers in between the labeled anchors. Higher scores indicate more severe symptoms, bother, or impact.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline